CLINICAL TRIAL: NCT05721001
Title: NEO - E-vita Open Neo Treatment of Aortic Arch Aneurysms and Dissections
Brief Title: French Registry Conducted on E-vita OPEN NEO
Acronym: NEO
Status: Active, not recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: NEO
Record Dates: First submitted 2023-01-06; First posted 2023-02-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Vascular Aneurysm
Keywords: Thoracic; Aorta; Aneurysm; Dissection; Open; Repair; Frozen; Elephant; Trunk
MeSH Terms: conditions — Aneurysm | interventions — Sutureless Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Surgical Repair — In Frozen Elephant Trunk procedure, the proximal aortic arch is replaced with a dacron graft, and a thoracic stent graft, sutured to the distal end of the dacron prosthesis, is deployed antegradely into the descending aorta. This mostly one-stage alternative approach eliminates the interval mortality rate related to the conventional elephant trunk procedure. Moreover, it constitutes a solution in fragile patients who cannot safely complete a second major operation after surviving the first.
  Other Names: Frozen Elephant Trunk Technique

SUMMARY:
Observational, prospective/retrospective, non-randomised, non-comparative, multicentre cohort study.

Primary objective is evaluation of in-hospital all-cause mortality after treatment of extensive acute and chronic aortic pathologies with E-vita OPEN NEO.

DETAILED DESCRIPTION:
Objectives

Primary objective:

• Evaluation of in-hospital all-cause mortality after treatment of extensive acute and chronic aortic pathologies with E-vita OPEN NEO

Secondary objective:

• Evaluation of the morbi-mortality in-hospital, 1 year and 3 years follow-up after treatment of extensive acute and chronic aortic pathologies with E-vita OPEN NEO.

Morbidity is defined as:

* new permanent (> 30 days) neurological complications (stroke mRS > 2, spinal cord ischemia, paraparesis, paraplegia)
* new clinical malperfusion (including visceral malperfusion)
* new permanent (>90 days) renal insufficiency requiring dialysis or hemofiltration in patients with normal pre-procedure serum creatinine level The others secondary objectives are to assess changes of the stent graft system in the medium (1 year) and long term (3 years):
* type Ib, II, or IV endoleaks in patients with aneurysm or type Ib or II entry flow in patients with dissection
* permeability of the vascular part

Patient population All patients treated with E-vita OPEN NEO until 31st March 2024 will be included in this registry if they are not opposed to the study. Follow-up of these patients will end in 2027.

Patients to be documented:

All male and female patients who have undergone implantation of E-vita OPEN NEO at their physician's discretion in France since device CE marking in 2020 and until 31st March 2024.

Inclusion/Exclusion Criteria None Indications for Use for E-vita OPEN NEO are listed in the device IFU. Patients are treated with E-vita OPEN NEO at the discretion of the treating physician.

Methodology In this study, we will conduct an observational cohort of consecutive patients who receive / received an E-vita OPEN NEO implant for the treatment of extensive acute or chronic aortic pathologies until 31st March, 2024. Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with E-vita OPEN NEO. All patients will be provided with a non-objection letter and given the opportunity to refuse to participate. Patients will either receive the non-objection letter before treatment or it is mailed to them by their treating physician.

A screening log will be kept during the study. In the screening log it will be documented which patients objected to the collection of their data and were therefore not included in the registry. The number of E-vita OPEN NEO implanted in France during the enrolment phase of the study will be submitted and compared to the number of patients enrolled in the study to assess the coverage of the study.

Patient data will be documented at the following time points: Pre-operative planning, intervention, prior to discharge from hospital, 1 year, and 3 years follow-up. The period of data collection will be 3 years ± 6 months (depending on the time point of the 3 years follow-up visit) starting from the intervention for each patient. All adverse events defined prior to study start will be adjudicated by the Clinical Event Committee (CEC).

Inclusion period (retrospective/prospective): Q3 2022 till Q1 2024 Follow-up: 3 years Total study period: 6 years

ELIGIBILITY:
Inclusion Criteria:

* non-objection from the patient for data collection within this Registry
* patient treated with E-vita Open NEO

Exclusion Criteria:

* objection from the patient for data collection within this Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All male and female patients who have undergone implantation of E-vita OPEN NEO at their physician's discretion in France since device CE marking in 2020 and until 31st March 2024 will receive a non-objection letter. If patient does not object to his/her data collection, patient will be enrolled and data collection can start.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 3 years
  Rate of in-hospital all-cause mortality

SECONDARY OUTCOMES:
Mortality | 1 year and 3 years
  All-cause mortality
Morbidity | 1 year and 3 year
  new neurological complication (defined as stroke, spinal cord ischemia, paraparesis, paraplegia), new clinical malperfusion (including visceral malperfusion), new permanent (> 90 days) renal insufficiency requiring dialysis or hemofiltration in patients with normal pre-procedure serum creatinine level
Severe Adverse Events | 1 year
  Rate of patients with SAE until 1 year follow-up (device-related, procedure-related, disease-related)
Severe Adverse Events | 3 years
  Rate of patients with SAE between 1 year and 3 year year follow-up (device-related, procedure-related, disease-related)
Neurological complications | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New permanent (> 30 days) neurological complications
Neurological complications | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New transient (≤ 30 days) neurological complications
Stroke | At discharge, an average of 45 days, 1 year, 3 years
  New permanent (> 30 days) stroke
Stroke | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New transient (≤ 30 days) stroke
Paraplegia | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New permanent (> 30 days) paraplegia
Paraparesis | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New permanent (> 30 days) paraparesis
Paraparesis | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New transient (≤ 30 days) paraparesis
Malperfusion | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New clinical visceral malperfusion
Renal Insufficiency | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New transient (≤ 90 days) renal insufficiency requiring dialysis or hemofiltration
Renal Insufficiency | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with New permanent (> 90 days) renal insufficiency requiring dialysis or hemofiltration
Permeability | 1 year, 3 years
  Rate of patients with Permeability of the vascular part
Reinterventions | 1 year, 3 years
  Rate of patients with Reinterventions (device-related, procedure-related, disease-related)
Additional interventions | 1 year, 3 year
  Rate of patients with Unplanned / planned additional interventions
Bleeding | At discharge, an average of 45 days, 1 year, 3 years
  Re-exploration due to bleeding
Endoleaks | At discharge, an average of 45 days, 1 year, 3 years
  Rate of patients with Endoleak type Ib, II, III or IV
False Lumen | At discharge, an average of 45 days, 1 year, 3 year
  Rate of patients with Obliterated, completely thrombosed, partially thrombosed, or patent false lumen in the stented region
Entry flow | At discharge, an average of 45 days, 1 year, 3 year
  Rate of patients with Type Ib, II or R entry flow, endoleak of unknown origin

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Fouquet, Prof, Principal Investigator — Centre Hospitalo-Universitaire d'Angers
Locations (23):
- France (23):
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalo-Universitaire d'Angers, Angers
  - Centre Hospitalier Annecy Genevois, Annecy
  - CHU Besançon, Besançon
  - Clinique Saint-Augustin, Bordeaux
  - Hôpital de La Cavale Blanche - Brest, Brest
  - Hôpital Louis PRADEL, Bron
  - Hôpital Privé Saint-Martin, Caen
  - Clinique de l'Infirmerie Protestante, Caluire-et-Cuire
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Chu Henri Mondor, Créteil
  - CHU le Bocage - CHU de Dijon, Dijon
  - Hôpital Privé Bois Bernard, Lens
  - CHU Lille, Lille
  - CHRU Limoges - Dupuytren, Limoges
  - CHU Montpellier, Montpellier
  - Groupe Hospitalier de la région de Mulhouse et Sud Alsace GHRMSA (Mulhouse), Mulhouse
  - APHP Pitié Salpétrière, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rennes - CHRU Pontchaillou, Rennes
  - CHU Rouen (Charles Nicolle), Rouen
  - Hopitaux Universtaires Strasbourg, Strasbourg
  - CHU de Tours - Hôpital Trousseau, Tours